CLINICAL TRIAL: NCT01402440
Title: An Open-Label, Single-arm, Phase I Study of AEB071 (a Protein Kinase C Inhibitor) in Patients With CD79-mutant Diffuse Large B-Cell Lymphoma
Brief Title: Study of AEB071 (a Protein Kinase C Inhibitor) in Patients With CD79-mutant Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to enrolment challenges and availability of other options for DLBCL patients. The termination is not a consequence of any safety concern.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COEB071X2101; 2010-024367-41 (EudraCT Number)
Record Dates: First submitted 2011-07-05; First posted 2011-07-26 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2015-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma,; Phase 1,; CD79 Mutation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — sotrastaurin

ARMS (1):
- AEB071 (Experimental)
  Interventions: Drug: AEB071

INTERVENTIONS:
Drug: AEB071

SUMMARY:
This study has two phases, a dose escalation phase and a dose expansion phase. For dose escalation, the primary objective is to estimate the maximum tolerated dose of AEB071 in patients with diffuse large b-cell lymphoma. The endpoint for this objective will be occurrence of Dose Limiting Toxicity. For dose expansion, the primary objective is to characterize the safety and tolerability of the maximum tolerated dose or recommended phase 2 dose of AEB071 in patients with diffuse large b-cell lymphoma. The endpoints for this objective will be occurrence of Adverse Events (AEs), Serious Adverse Events (SAEs), assessment of clinical laboratory values, and vital sign measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse large B-cell lymphoma (DLBCL) with activating mutations in CD79 (A or B subunits). DLBCL that arose from transformed indolent lymphoma is allowed.
* Prior treatment and relapse following anthracycline-based chemotherapy and autologous bone marrow or stem cell transplant. Patients who are not transplant eligible may be considered for the study following a single regimen of chemotherapy such as R-CHOP or R-EPOCH alone. There is no limit to prior therapy allowed.

  * Patients may be treated with localized radiation to as many as two sites of disease, so long as measurable or evaluable disease remains at untreated sites.
  * Patients may be treated with corticosteriods immediately prior to enrollment and during the course of the study treatment as long as steriod treatment is tapered to a toal daily dosage of 10mg or less of prednisone (or it's equivalent) prior to AEB071 administration
* WHO performance status of ≤2

Exclusion Criteria:

* Patients at screening who are treated with strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) that can not be discontinued.
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:
* History or presence of ventricular tachyarrhythmia
* Presence of unstable atrial fibrillation (ventricular response > 100 bpm); Patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria.
* Angina pectoris or acute myocardial infarction ≤ 3 months prior to starting study drug
* Other clinically significant heart disease (e.g., symptomatic congestive heart failure; uncontrolled arrhythmia or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen)
* Patients with another malignancy that was treated within the last three years with the exceptions of localized basal cell carcinoma and cervical carcinoma.
* Patients with impairment of GI function or GI disease that could interfere with the absorption of AEB071.
* Patients with a known history of Human Immunodeficiency Virus (HIV)

  * HIV testing is not required as part of this study
* Patients with a known history of active hepatitis B or C infection unless they are on antiviral therapy

  * The determination of active hepatitis status should be as per standard of care at each site
  * Hepatitis B and C testing is not required as part of this study

Time since the last prior therapy for treatment of underlying malignancy**:

* Cytotoxic chemotherapy: ≤ than the duration of the most recent cycle of the previous regimen (with a minimum of 2 weeks for all)
* Biologic therapy (e.g., antibodies): ≤ 4 weeks
* ≤ 5 x t1/2 of a small molecule therapeutic, not otherwise defined above

  **Patients must have recovered or stabilized from all toxicities related to their previous treatment except for alopecia
* Patients with any history of significant coagulopathy or a medical condition requiring long term systemic anticoagulation that would interfere with biopsies.
* Patients having undergone major surgery less than 4 weeks prior to enrollment or that have not fully recovered from prior surgery.
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Frequency of Dose Limiting Toxicity (DLT) during cycle 1 (Dose Escalation phase) | Cycle 1 (28 days)
Number of Pparticipants reporting Serious Adverse Events and Adverse Events (Dose Expansion phase) | Baseline, 28 days

SECONDARY OUTCOMES:
Overall Response Rate, using NHLIWG criteria | Baseline, 12 months
  Assess the overall response rate to AEB071
Number of Participants reporting Serious Adverse Events and Adverse Events | Baseline, 12 months
AEB071 PK parameters including Cmax, tmax, AUCt, Ctrough, CL/F and RA | First 7 months of treatment period
  Evaluate the single and multiple dose PK of AEB071 in patients with Diffuse Large B-Cell Lymphoma (DLBCL)
Pre and post-dose gene and protein expression of cytokines and any correlations with exposure to AEB071 | First 7 months of treatment period
  Assess the pharmacodynamic response to AEB071 in Lymphoma and blood specimens

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novarts Pharmaceuticals, Study Director — Novarts Pharmaceuticals
Locations (23):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Washington University School of Medicine Div. of Medical Oncology, St Louis, Missouri
  - Hackensack University Medical Center Hackensack (SC), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center MSK 2, New York, New York
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital Ohio State, Columbus, Ohio
  - University of Texas/MD Anderson Cancer Center SC Location, Houston, Texas
- France (4):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pierre-Benite Cédex
  - Novartis Investigative Site, Rouen
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, München
- Novartis Investigative Site, Shatin, New Territories, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Torino, TO
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Manchester, United Kingdom

REFERENCES:
- See also: Results for OEB071X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13343